CLINICAL TRIAL: NCT06412211
Title: Clinical Utility of Photoacoustic Finder in Sentinel Lymph Node Detection in Breast Cancer - Pilot Study
Brief Title: A Clinical Feasibility Study of a Photoacoustic Finder
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Pohang University of Science and Technology (Other)
Responsible Party: Principal Investigator, Dooreh Kim, Clinical Assistant Professor, Seoul St. Mary's Hospital
Other Study IDs: KC21DIDT0810
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Sentinel Lymph Node; Breast Cancer
Keywords: Photoacoustic; Sentinel lymph node detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SLN resected patients: Patients with breast cancer underwent sentinel lymph node biopsy
  Interventions: Device: Photoacoustic finder

INTERVENTIONS:
Device: Photoacoustic finder — Sentinel lymph node detector using photoacoustic signal

SUMMARY:
Determining the prognosis of breast cancer relies significantly on axillary staging by sentinel lymph node biopsy (SLNb). The SLNb is generally performed using radioisotopes, blue dyes, or both to improve the false negative rate. However, a gamma probe with radioisotopes involves ionizing radiation, and blue dye detection relies on visual inspection by an operator. To overcome these limitations, the photoacoustic finder (PAF) was developed as a highly sensitive, non-radioactive detector that uses only blue dye and a photoacoustic signal to detect SLNs. To evaluate the PAF, its performance was compared with the standard SLN detection method for breast cancer patients.

DETAILED DESCRIPTION:
-Introduction The presence of lymphatic metastases in breast cancer patients is an important prognostic factor for survival, and accurate staging leads to appropriate adjuvant treatment. Sentinel lymph node biopsy (SLNb) is a standard method used to confirm regional axillary lymphatic metastases in breast cancer patients. Sentinel lymph nodes (SLNs) are a group of initial lymph nodes (LNs) located in proximity to the tumor and connected via lymphatic vessels (LVs), hypothetically the first ones that a primary tumor drains in the regional lymphatic basin. If metastatic tumor cells are not confirmed in the excised SLNs, the incidence of morbidities, such as lymphedema, can be reduced by omitting unnecessary axillary lymph node dissection (ALND). The SLNb procedure is a dual-modal method utilizing a radioactive tracer (e.g., 99mTc) and/or blue dye to identify the SLNs. The radioactive tracer and blue dye are administered before surgery and absorbed by the lymphatic system, and eventually they flow into the SLNs. During the surgical procedures, the SLNs are identified through visual inspection of blue-dyed LVs and radioactivity detection using a gamma probe. The identified SLNs are subsequently excised and sent for pathological examination to assess the potential metastatic tumor.

The dual-modal method enhances the accuracy and efficiency of SLN identification by leveraging the distinct advantages of each method. However, the radioactive isotopes in the SLNb surgery present an inherent radiation exposure risk and necessitate specialized facilities and skilled medical personnel. These factors introduce complexities into the surgical procedure and create obstacles for the implementation of SLNb in local hospitals. Moreover, the administration of radioactive material typically requires cooperation with a nuclear medicine department, which restricts direct usage by the surgeon and may impact surgical scheduling. Lastly, because radioactive isotopes do not provide visual information, the intuitive identification of SLNs is challenging. On the other hand, blue dye visually stains the lymphatic network, enabling the intuitive identification of SLNs without radiation exposure. However, relying on visual inspection of blue-dyed SLNs may introduce inter-physician variability and potential inaccuracies in identifying SLNs, owing to variable lesion characteristics such as the presence of adipose tissue and blood. These limitations make it challenging to see blue dye within LNs, ultimately leading to reduced sensitivity in the SLN detection.

Photoacoustic (PA) imaging or sensing is a non-ionizing technique that utilizes the intrinsic light absorption properties of biological tissue components . To generate PA signals, a nanosecond pulsed laser induces repeated instantaneous thermal expansions within a sample, creating acoustic waves . These acoustic waves are then captured by an ultrasound transducer and analyzed to confirm the presence of specific constituents within the sample. PA sensing technology can detect dye-stained LNs with high sensitivity and provide a real-time quantitative representation. This method can precisely determine the presence or absence of dyed SLNs that may have been indistinguishable through visual inspection. Consequently, it can facilitate SLNb procedures without radioactive materials. In our previous studies, a cutting-edge system known as the photoacoustic finder (PAF) was successfully deviesed. It is remarkably efficacious in detecting SLNs while maintaining a high signal-to-noise ratio (SNR). The PAF combines a solid-state dye (SSD) laser handpiece and a transparent ultrasound transducer (TUT) in a precisely coaxial configuration. This study describes preclinical trials of the PAF, which confirmed its ability to accurately detect blue-dyed SLNs.

This cross-sectional clinical study was conducted ex vivo to validate the feasibility of using the PAF in a clinical setting. The process confirms the signal from excised LNs identified by the dual-modal method and the PAF before sending them to pathology. To determine its detection performance, the effectiveness of PAF is compared to the detection rate of standard SLNb. The results establish the clinical feasibility of using PAF for SLNb, providing a non-radioactive alternative.

-Study design: This study was conducted as a cross-sectional, open-label, single-arm ex vivo study within a single institution to investigate the efficacy of PAF compared to standard dual-modal methods for SLN detection in the treatment of breast cancer. The SLNb procedures followed international guidelines, using both radioisotope and blue dye mapping. SLNs were identified using gamma probe and blue dye visual inspection, then resected and labeled to reconfirm the with gamma probe and blue dye visual inspection. Subsequently, PAF was employed to capture signals from the LNs. To minimize potential errors such as labeling mistakes and LN delivery errors, the PAF system was placed in the operating room. The study enrolled women diagnosed with breast cancer who presented to the Department of Breast Surgery at St. Mary's Hospital, Seoul, The Republic of Korea.

-Sentinel lymphnode biopsy: The SLNb was performed in accordance with established international guidelines, utilizing both radioisotope and blue dye mapping methods. Five surgical oncologists participated in the study, all of whom were experienced in performing standard dual-modal SLNb and understood the clinical protocol. The radioisotope (0.1 mL of 99mTc-phytate) was administered into the subdermal lymphatic flexus under the areola within 30 minutes to 8 hours prior to operation. When the surgery started, the operator confirmed the location of the tumor. Then, a blue dye (indigo carmine, 2-5 ml) was injected peritumorally or periareolarly prior to incision, with subsequent massaging for 1 minute following injection. The axillary nodal basin was closely examined using a handheld gamma probe to detect radioactive signals and visually examined by the naked eye to detect grossly blue-dyed LNs. The identification of SLNs continued until either no further signal was detected by the gamma probe or blue-dyed LNs were no longer found in the nodal basins within the operation field. For this study, SLNs were defined as LNs with a gamma probe signal greater than 10% of the maximum signal value and/or visibly stained with blue dye. Additionally, based on the surgeon's experience, abnormally palpable LNs that were not detected by gamma probe and visual inspection were also excised, and these were labeled as non-SLNs. The SLNs and non-SLNs were further examined by PAF, and subsequently were forwarded to the pathology department for frozen section analysis.

-Sample Size: To determine the required sample size for testing the non-inferiority of PAF and the dual-modal method, the non-inferiority chi-square sample size estimator was utilized, employing a non-inferiority margin of 5%, a significance level (alpha) of 5%, and a power (1-beta) of 80%. Drawing from prior research and based on experimental data from tests, it was assumed that the visual detection rate would be approximately 78% for SLNs and 84% for PAF. Calculations revealed that a total of 157 SLNs would be necessary, corresponding to approximately 1.5 SLNs per patient, thus requiring the enrollment of 115 patients to fulfill the sample size requirements with an anticipated 10% drop-out.

-Static Analysis Methods:

The primary endpoints, which were the SLN detection rates for the gamma probe, visual inspection, and PAF were defined as follows:

Detection rate= (Number of detected SLNs)/(Total number of SLNs) ×100 [%]

The secondary endpoints encompassed the results of a non-inferiority analysis conducted using the chi-square test. Additionally, the sensitivity and specificity were assessed through ROC curve analysis as part of the additional endpoints. Regarding primary and secondary endpoints, SLNs were specifically examined, excluding non-SLNs to minimize potential surgeon subjectivity.

The Wilcoxon Mann-Whitney U-Test was performed to determine the cutoff for the PAF, and the statistical significances between 99mTc+/-, blue+/-, and non-injected groups were compared. In a non-inferiority analysis, a chi-square test was performed to compare the risk differences for 99mTc+, blue+, and PAF+ nodes. The independent samples t-test was used for other normal distributions, such as age and BMI. All statistical analyses in this study were conducted using MATLAB R2022a with the Statistics and Machine Learning Toolbox.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 74 years
* histologically confirmed invasive breast cancer or intraepithelial carcinoma
* no clinical suspicion of axillary LN metastasis

Exclusion Criteria:

* Previously undergone ipsilateral breast
* Axillary surgery
* Received chemotherapy prior to surgery
* who were unable to undergo SLN biopsy
* who had confirmed axillary LN metastasis by histologic examination
* who had breast cancer while lactating or pregnant

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A woman is diagnosed with breast cancer at St Mary's Hospital, Seoul.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Sentinel lymph node detection (SLN) rate | during the surgery
  Number of detected SLNs / Number of total resected LNs

CONTACTS AND LOCATIONS:
Overall Officials: Dooreh Kim, MD, Study Chair — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Provide clinical metrics and PAF signals for individual participant data.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Receive the data request via the registered email, verify the identity (for example, Relevant researcher), and provide the data.

REFERENCES:
- [Background] Kherlopian AR, Song T, Duan Q, Neimark MA, Po MJ, Gohagan JK, Laine AF. A review of imaging techniques for systems biology. BMC Syst Biol. 2008 Aug 12;2:74. doi: 10.1186/1752-0509-2-74. PMID 18700030
- [Background] Stoffels I, Jansen P, Petri M, Goerdt L, Brinker TJ, Griewank KG, Poeppel TD, Schadendorf D, Klode J. Assessment of Nonradioactive Multispectral Optoacoustic Tomographic Imaging With Conventional Lymphoscintigraphic Imaging for Sentinel Lymph Node Biopsy in Melanoma. JAMA Netw Open. 2019 Aug 2;2(8):e199020. doi: 10.1001/jamanetworkopen.2019.9020. PMID 31411710
- [Background] Kim C, Song KH, Gao F, Wang LV. Sentinel lymph nodes and lymphatic vessels: noninvasive dual-modality in vivo mapping by using indocyanine green in rats--volumetric spectroscopic photoacoustic imaging and planar fluorescence imaging. Radiology. 2010 May;255(2):442-50. doi: 10.1148/radiol.10090281. PMID 20413757
- [Background] Hudis CA, Barlow WE, Costantino JP, Gray RJ, Pritchard KI, Chapman JA, Sparano JA, Hunsberger S, Enos RA, Gelber RD, Zujewski JA. Proposal for standardized definitions for efficacy end points in adjuvant breast cancer trials: the STEEP system. J Clin Oncol. 2007 May 20;25(15):2127-32. doi: 10.1200/JCO.2006.10.3523. PMID 17513820
- [Background] Krag DN, Anderson SJ, Julian TB, Brown AM, Harlow SP, Costantino JP, Ashikaga T, Weaver DL, Mamounas EP, Jalovec LM, Frazier TG, Noyes RD, Robidoux A, Scarth HM, Wolmark N. Sentinel-lymph-node resection compared with conventional axillary-lymph-node dissection in clinically node-negative patients with breast cancer: overall survival findings from the NSABP B-32 randomised phase 3 trial. Lancet Oncol. 2010 Oct;11(10):927-33. doi: 10.1016/S1470-2045(10)70207-2. PMID 20863759
- [Background] Petrelli F, Lonati V, Barni S. Axillary dissection compared to sentinel node biopsy for the treatment of pathologically node-negative breast cancer: a meta-analysis of four randomized trials with long-term follow up. Oncol Rev. 2012 Oct 8;6(2):e20. doi: 10.4081/oncol.2012.e20. eCollection 2012 Oct 2. PMID 25992218
- [Background] Naik AM, Fey J, Gemignani M, Heerdt A, Montgomery L, Petrek J, Port E, Sacchini V, Sclafani L, VanZee K, Wagman R, Borgen PI, Cody HS 3rd. The risk of axillary relapse after sentinel lymph node biopsy for breast cancer is comparable with that of axillary lymph node dissection: a follow-up study of 4008 procedures. Ann Surg. 2004 Sep;240(3):462-8; discussion 468-71. doi: 10.1097/01.sla.0000137130.23530.19. PMID 15319717
- [Background] Veronesi U, Paganelli G, Viale G, Luini A, Zurrida S, Galimberti V, Intra M, Veronesi P, Maisonneuve P, Gatti G, Mazzarol G, De Cicco C, Manfredi G, Fernandez JR. Sentinel-lymph-node biopsy as a staging procedure in breast cancer: update of a randomised controlled study. Lancet Oncol. 2006 Dec;7(12):983-90. doi: 10.1016/S1470-2045(06)70947-0. PMID 17138219
- [Background] Kim T, Giuliano AE, Lyman GH. Lymphatic mapping and sentinel lymph node biopsy in early-stage breast carcinoma: a metaanalysis. Cancer. 2006 Jan 1;106(1):4-16. doi: 10.1002/cncr.21568. PMID 16329134
- [Background] Krag D, Weaver D, Ashikaga T, Moffat F, Klimberg VS, Shriver C, Feldman S, Kusminsky R, Gadd M, Kuhn J, Harlow S, Beitsch P. The sentinel node in breast cancer--a multicenter validation study. N Engl J Med. 1998 Oct 1;339(14):941-6. doi: 10.1056/NEJM199810013391401. PMID 9753708
- [Background] Pesek S, Ashikaga T, Krag LE, Krag D. The false-negative rate of sentinel node biopsy in patients with breast cancer: a meta-analysis. World J Surg. 2012 Sep;36(9):2239-51. doi: 10.1007/s00268-012-1623-z. PMID 22569745
- [Background] Wang Z, Wu LC, Chen JQ. Sentinel lymph node biopsy compared with axillary lymph node dissection in early breast cancer: a meta-analysis. Breast Cancer Res Treat. 2011 Oct;129(3):675-89. doi: 10.1007/s10549-011-1665-1. Epub 2011 Jul 9. PMID 21743996
- [Background] Park B, Han M, Park J, Kim T, Ryu H, Seo Y, Kim WJ, Kim HH, Kim C. A photoacoustic finder fully integrated with a solid-state dye laser and transparent ultrasound transducer. Photoacoustics. 2021 Aug 4;23:100290. doi: 10.1016/j.pacs.2021.100290. eCollection 2021 Sep. PMID 34401325